CLINICAL TRIAL: NCT07005544
Title: Improving Hand Hygiene Skills Using Virtual Reality: A Quasi-Experimental Approach
Brief Title: Hand Hygiene Skills Using Virtual Reality
Acronym: RealityCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RealityCare TED 2021-130383B-I
Record Dates: First submitted 2025-05-23; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Virtual Reality; Hand Washing Behavior
Keywords: Virtual Reality; Infection Control; Hand Hygiene; Caregivers

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, one-group pretest-posttest study evaluated the effectiveness of a Virtual Reality hand hygiene training program for auxiliary nurses and informal caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Handwashing using virtual reality
  Interventions: Device: RealityCare

INTERVENTIONS:
Device: RealityCare — Participants utilized a Virtual Reality scenario that simulated a complete handwashing sequence with water and soap, including an instructional display demonstrating the correct hand hygiene technique.

SUMMARY:
Quasi-experimental, one-group pretest-posttest study evaluated the effectiveness of a Virtual Reality hand hygiene training program for auxiliary nurses and informal caregivers in Colombia

DETAILED DESCRIPTION:
This quasi-experimental, one-group pretest-posttest study evaluated the effectiveness of a Virtual Reality hand hygiene training program for auxiliary nurses and informal caregivers in Colombia. A total of 215 participants (94 auxiliary nurses, 121 informal caregivers) completed the intervention, which included three 15-minute Virtual Reality training sessions with real-time feedback on hand hygiene technique. Data were collected at baseline (PRE) and immediately after the Virtual Reality intervention (POST), which included one 15-minute training sessions. Variables assessed included hand hygiene performance, error rates, and knowledge assessment. Linear mixed-effects models were used to assess changes over time.

ELIGIBILITY:
Inclusion Criteria:

* auxiliary nurses,
* informal caregivers

Exclusion Criteria:

- Caregivers (both auxiliary nurses or informal caregivers) with prior healthcare training or experience with virtual reality were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Errors | From baseline to the end of treatment on the same day, within an estimated period of 1 to 2 hours
  Number of errors based on the standardized hand hygiene protocol approved by institutions involved in this study
Time | From baseline to the end of treatment on the same day, within an estimated period of 1 to 2 hours
  Time (measure in seconds) used for washing the hands

SECONDARY OUTCOMES:
Knowledge | From baseline to the end of treatment on the same day, within an estimated period of 1 to 2 hours
  Number of right responses to key questions about hand hygiene

CONTACTS AND LOCATIONS:
Overall Officials: Jose Mira, PhD, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Universidad Minuto de Dios, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
Anonymized data are analyzed by FISABIO

REFERENCES:
- [Background] Stuart JP, Gannon PR, Dotto VR, Regina R, Mumma JM. Visualizing the WHO "My Five Moments for Hand Hygiene," framework: A virtual reality training program for improving hand hygiene adherence among nurses. Am J Infect Control. 2025 May;53(5):576-581. doi: 10.1016/j.ajic.2025.01.007. Epub 2025 Jan 15. PMID 39824286
- [Background] Omori K, Shigemoto N, Kitagawa H, Nomura T, Kaiki Y, Miyaji K, Akita T, Kobayashi T, Hattori M, Hasunuma N, Tanaka J, Ohge H. Virtual reality as a learning tool for improving infection control procedures. Am J Infect Control. 2023 Feb;51(2):129-134. doi: 10.1016/j.ajic.2022.05.023. Epub 2022 Jun 1. PMID 35659561
- [Background] Eichel VM, Brandt C, Brandt J, Jabs JM, Mutters NT. Is virtual reality suitable for hand hygiene training in health care workers? Evaluating an application for acceptability and effectiveness. Antimicrob Resist Infect Control. 2022 Jun 25;11(1):91. doi: 10.1186/s13756-022-01127-6. PMID 35752839
- [Derived] Mira J, Gonzalez M, Villalba C, Guerra L, Ramirez-Moya Y, Hernandez J, Moya O, Pineda L, Perez-Esteve C. Improving Hand Hygiene Skills Using Virtual Reality: Quasi-Experimental Study. J Med Internet Res. 2025 Oct 7;27:e78882. doi: 10.2196/78882. PMID 41057041
- See also: Training informal caregivers using virtual reality to increase patient safety — https://realitycare.es